CLINICAL TRIAL: NCT00357318
Title: A Phase I Study of Bevacizumab in Combination With SU11248
Brief Title: Bevacizumab and Sunitinib in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00185; NCI-2009-00185 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000489184; CASE 5Y05 (Other: Case Comprehensive Cancer Center); 7537 (Other: CTEP); P30CA043703 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Sunitinib; Bevacizumab

ARMS (1):
- Treatment (sunitinib malate, bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29 and oral sunitinib malate (SU11248) once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Biological: bevacizumab; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of bevacizumab and sunitinib in treating patients with solid tumors. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and sunitinib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving bevacizumab together with sunitinib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of bevacizumab in combination with sunitinib malate (SU11248) in patients with solid tumors.

SECONDARY OBJECTIVES:

I. Evaluate the objective response rate, time to disease progression, and overall survival of these patients.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29 and oral sunitinib malate (SU11248) once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bevacizumab and SU11248 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 10 patients are treated at the MTD.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic/unresectable adrenocortical carcinoma or melanoma not amenable to curative surgical or radiation therapy.
* Accrual closed as of 5/27/2009 to patients with renal cell carcinoma
* No squamous cell histology
* No histology in close proximity to a major blood vessel
* No history of or known brain metastases, spinal cord compression, or carcinomatous meningitis
* No new evidence of brain or leptomeningeal disease on screening CT scan or MRI
* ECOG performance status (PS) 0-1 OR Karnofsky PS 60-100%
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥100,000/mm³
* Hemoglobin ≥ 10.0 g/dL
* Calcium ≤ 12.0 mg/dL
* Urine protein:creatinine ratio ≤ 0.5 by urinalysis
* Patients with urine protein:creatinine ratio > 0.5 must have proteinuria < 1,000 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* None of the following within the past 12 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Severe peripheral vascular disease (claudication) or procedure on peripheral vasculature
  * Coronary/peripheral artery bypass graft
  * New York Heart Association (NYHA) grade III-IV congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Clinically significant bleeding
  * Deep venous thrombosis
  * Pulmonary embolism
  * No ongoing cardiac dysrhythmias of NCI CTCAE ≥ grade 2, atrial fibrillation of any grade, or prolongation of the QTc interval to > 450 msec (males) or > 470 msec (females)
  * No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
  * No condition classified as NYHA grade III or IV
  * No hypertension that cannot be controlled by medications
  * Blood pressure < 140/90 mm Hg
  * No evidence of bleeding diathesis or coagulopathy
  * No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * No history of or known brain metastases, spinal cord compression or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening CT or MRI scan unless without progression on * MRI or CT for 3 months."
  * No significant traumatic injury within the past 28 days
  * No serious, non-healing wound, ulcer, or bone fracture
  * No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
  * No known HIV or AIDS-related illness
  * No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation.
* Recovered from prior radiation therapy, surgery, or other prior therapy
* No prior bevacizumab or sunitinib malate (SU11248)
* Other antiangiogenic therapies allowed
* No prior tyrosine kinase inhibitor of the VEGF receptor or bevacizumab for patients with metastatic renal cell carcinoma
* No major surgical procedures or open biopsy within the past 28 days
* No core biopsy within the past 7 days
* No radiation therapy or systemic therapy within the past 4 weeks
* No concurrent full-dose anticoagulants (e.g., warfarin)
* Concurrent low-dose anticoagulation (e.g., prophylactic port patency) allowed
* No concurrent treatment on another clinical trial
* No other concurrent investigational drugs
* No concurrent major surgery
* No other concurrent anticancer agents or therapies, including chemotherapy, biological response modifiers, hormonal therapy, surgery, palliative radiation therapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bevacizumab in combination with sunitinib malate determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | 42 days

SECONDARY OUTCOMES:
Objective response rate assessed by RECIST | Up to 5 years
Overall survival | Up to 5 years
  Will be summarized using the method of Kaplan and Meier. 95% confidence intervals will be reported when appropriate.
Progression-free survival | Up to 5 years
  Will be summarized using the method of Kaplan and Meier. 95% confidence intervals will be reported when appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio